CLINICAL TRIAL: NCT07033013
Title: A Randomized, Double Blind, Placebo Controlled, Clinical Study to Examine the Benefits of an Oral Product in Panelists With Menopausal Symptoms Including Vasomotor Symptoms (VMS).
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olly, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UNLV20250320
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Instructions: Take 1 capsule when having a hot flash at the onset of a hot flash (not to exceed 1 capsule/day). Only treat 1 hot flash during a 24-hour period.
  Interventions: Dietary Supplement: Placebo
- Dietary Supplement with actives (Active Comparator): Instructions: Take 1 capsule when having a hot flash at the onset of a hot flash (not to exceed 1 capsule/day). Only treat 1 hot flash during a 24-hour period.
  Interventions: Dietary Supplement: Dietary Supplement with actives

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Dietary Supplement with actives — Dietary supplement containing EstroG-100 and GABA
  Arms: Dietary Supplement with actives

SUMMARY:
Randomized, Double-Blind, Placebo-Controlled, Single-Center Clinical Study with a Run-in Baseline, Daily Diary Log, and Validated Questionnaires (Greene GCS) with Oral Dietary Supplement

ELIGIBILITY:
Inclusion Criteria:

* Healthy Females aged 40 to 65 years
* Self-reporting menopausal symptoms (> 5 hot flashes per day) and have been present for a minimum of previous 60 days prior to baseline visit
* Reporting a variable cycle length of > 7 days different from normal
* NORMAL BMI (per metropolitan life tables): under 30 kg/m2
* Able to read, understand, and complete the study questionnaire and records.
* Able to understand the study procedures.
* Able to comply with all study requirements.
* Written informed consent to participate in the study.
* Willingness to actively participate in the study and to come to the scheduled visits.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Immune insufficiency
* Women of childbearing potential including those still having a menstrual cycle on a regular basis who are not perimenopausal, menopausal or post-menopausal.
* History of hysterectomy
* Women on hormone replacement therapy
* Use of systemic corticosteroids or immunosuppressant drugs.
* Other diseases or medications that might directly interfere in the study or put the panelist's health under risk, such as: thyroid disease, diabetes mellitus, history of hormone dependent (gynecological) cancer, endometrial hyperplasia, uterine cancer, endometrial cancer, drug and alcohol abuse, mental disorder, abnormality in renal and liver functions, personal or family history of breast cancer in a first degree relative, and history of clotting disorder such as deep vein thrombosis.)
* Cardiovascular, chronic liver, thyroid or kidney diseases; a history of cancer; a disease or condition that could influence the participants' ability to follow the study protocol
* Alcohol or drug abuse
* Use of hormonal contraceptives within the last 3 months
* Use of other menopause supplements or drugs
* Uncontrolled hypertension (160/100 mmHg or higher, measured after 10 min of seated rest)
* Oophorectomy or amenorrhea > two years.
* Participating in a different clinical trial within one month of the start of this clinical trial or planning to participate in another clinical trial during the trial period
* Continuous intake of foods based on Cynanchum wilfordii Hemsley, Phlomis umbrosa Turczaninow, and Angelica gigas Nakai within the past month
* Employees of the institute or the brand owner or the manufacturers of the product
* Note: Habitual medicine and supplement intake will be registered prior to inclusion in the study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
24 hour effects following single dose of Mellow Menopause - Hot Flashes | From baseline Day 7 to Treatement Day 1 (Day 8 of study)
  To assess the efficacy for improvement of a treatment product on menopausal vasomotor symptoms (hot flashes- intensity, duration) within 24 hours compared to placebo through daily diary data and MenoLife application based diary.

SECONDARY OUTCOMES:
Improvement of overall daily menopausal vasomotor symptoms | from enrollment to end of study at Day 15
  To assess the efficacy for improvement of overall daily menopausal vasomotor symptoms compared to placebo through daily diary data and MenoLife diary though 7 days. Data in the Daily diary and MenoLife Diary will be compared between the active supplement and placebo groups across different time points.

OTHER OUTCOMES:
Assess Menopause symptoms using the Greene Climacteric Scale (GCS). | from enrollment to end of study at Day 15
  To assess the efficacy of the investigation product on menopause symptoms using a validated questionnaire Greene Climacteric Scale (GCS). Data from the GCS Score will be compared between the active supplement and placebo groups across different time points.

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States